CLINICAL TRIAL: NCT01395459
Title: A Sustainable Approach to Increasing Cancer Screening
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Emmons, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15622; R01CA126596 (NIH)
Record Dates: First submitted 2011-07-09; First posted 2011-07-15 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer; Breast Cancer; Cervical Cancer
Keywords: screening; cancer prevention; IVR
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): Care as usual is given.
- IVR only (Experimental): The participants in this study arm receive calls from an Interactive Voice Response (IVR) call system, to remind them that they are in need of breast, cervical and colon cancer screening, as applicable.
  Interventions: Behavioral: IVR only
- IVR+PCC (Experimental): The participants in this study arm receive calls from an Interactive Voice Response (IVR) call system, to remind them that they are in need of breast, cervical and colon cancer screening, as applicable. Furthermore, if remained unscreened, these participants receive person to person follow up telephone calls from a prevention care coordinator (PCC) to address barriers.
  Interventions: Behavioral: IVR+PCC

INTERVENTIONS:
Behavioral: IVR only — As noted, patients in this arm receive consistent, but spaced out calls generated by an interactive voice response system reminding them of breast, cervical and colon cancer screenings needed, as applicable.
  Arms: IVR only
Behavioral: IVR+PCC — Interactive voice response calls followed up by prevention care coordinator calls for those who do not respond to IVR
  Arms: IVR+PCC

SUMMARY:
Parent study:

A Coordinated Approach to Cancer and Health (CATCH), was designed to compare the efficacy of two intervention arms (described below) intended to increase breast, cervical, and colon cancer screening rates among patients served by community health centers. A central focus of CATCH is to evaluate sustainable strategies for maximizing cancer screening rates among populations facing significant cancer disparities.

CATCH was conducted in partnership with the large health clinic in Massachusetts, which serves a largely Hispanic low income population. Focusing on the use of an Interactive Voice Response (IVR) telephone technology system, the study is examining the extent to which the IVR, when developed in a culturally sensitive and appropriate manner (focus groups will be conducted to inform the intervention), can improve breast, cervical and colon cancer screening rates compared to a control group. Furthermore, we plan to determine if pairing IVR with telephone calls from a prevention care coordinator (PCC) will result in higher screening rates (when compared to the IVR only group). We will determine the cost-effectiveness of IVR alone vs. IVR + PCC.

Substudy:

We conducted a substudy of the parent study, looking at a comparison of return rates of two colorectal cancer screening home test kits: Fecal Occult Bood Tests (gFOBTs) and Fecal Immunochemical Tests (FITs). As well we surveyed people who pick up one of these two types of tests to assess barriers and facilitators of returning the completed kit to the health center for assessment.

DETAILED DESCRIPTION:
For the substudy, the study objective was to:

Determine if there is a difference in completion of a home blood stool test kit by type of home test being employed Fecal Occult Blood Test (gFOBT) vs. Fecal Immunochemical Test (FIT), and to determine predictors of test completion.

Substudy methods/design/arms/eligibility:

All patients who picked up a home blood stool test kit during the 6-12 month study recruitment time period were randomized to receive either a gFOBT or FIT kit. Randomization occurred by the month. Medical assistants (MAs) handed out the kits. Participants who picked up a kit (either gFOBT or FIT) were given a study information card that briefly described the study and had a study opt out phone number on it. If patients did not call and opt out, the card let the patient know that he/she would be contacted via telephone to complete a brief survey, for which they were given a small incentive upon completion.

A bilingual member of the study staff telephoned individuals, who had not opted out, who picked up a home blood stool test kit during the study period. Four to six weeks post kit pickup, staff determined if the patient had returned a completed test to the clinic (yes vs. no) by examining the electronic medical record. This information- whether a patient had/had not returned a completed test was used to tailor some questions asked on the survey. Study staff obtained verbal informed consent before survey administration. Participants who cited that time was a burden stopping them from starting the survey were offered an abbreviated version of the survey.

This study was limited to age eligible patients who picked up a home colon cancer screening kit.

ELIGIBILITY:
Parent study only (please see detailed description for substudy)

Inclusion criteria

* All age and gender eligible patients, using GLFHC's guidelines, in need of: breast, cervical or colorectal cancer screenings.

Exclusion criteria

* All GLFHC patients who do are not age or gender eligible for a breast, cervical or colorectal cancer screening.

Substudy only: Inclusion: age eligible clinic patients who pick up either a gFOBT or FIT kit during the study period. Exclusion: non-age eligible patients who pick up a home test kit.

Ages: 21 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13675 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in population level cancer screening level at the health clinics involved. | year 3 of the study
  The primary outcome of interest is improvement of population-level screening and individual outcomes for 3 cancers (breast, cervical, and colorectal)of patients reached during the intervention.

OTHER OUTCOMES:
For the substudy: return rate of gFOBT kits vs. FITs | starting 4-6 weeks post pick up
  We are looking at return rates of 2 home colorectal cancer screening tests (gFOBT vs. FIT). We are contacting all people who picked up a kit to assess facilitators and barriers to return.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Emmons, PhD, Principal Investigator — Dana-Farber Cancer Institution
Locations (1):
- Greater Lawrence Family Health Center (GLFHC), Lawrence, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emmons KM, Cleghorn D, Tellez T, Greaney ML, Sprunck KM, Bastani R, Battaglia T, Michaelson JS, Puleo E. Prevalence and implications of multiple cancer screening needs among Hispanic community health center patients. Cancer Causes Control. 2011 Sep;22(9):1343-9. doi: 10.1007/s10552-011-9807-7. Epub 2011 Jul 5. PMID 21728056
- [Background] Greaney ML, De Jesus M, Sprunck-Harrild KM, Tellez T, Bastani R, Battaglia TA, Michaelson JS, Emmons KM. Designing audience-centered interactive voice response messages to promote cancer screenings among low-income Latinas. Prev Chronic Dis. 2014 Mar 13;11:E40. doi: 10.5888/pcd11.130213. PMID 24625364